CLINICAL TRIAL: NCT06836882
Title: The Effect of Sodium Hypochlorite and Chlorhexidine as Cavity Disinfectants on the Post Operative Pain and Success of Partial Caries Removal in Deep Carious Lesion With Moderate Pulpitis in Permanent Teeth: A Randomized Controlled Trial
Brief Title: Effect of Cavity Disinfectants on Post Operative Pain & Success of Partial Caries Removal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: shweta mittal
Record Dates: First submitted 2025-01-09; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Pulp Disease, Dental
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pt receiving SCR treatment (Active Comparator): No disinfectant solution was applied (control group).
  Interventions: Procedure: Selective caries removal
- Pt receiving SCR followed by disinfection with NaOCl (Experimental): the cavity was disinfected with 2.5% sodium hypochlorite
  Interventions: Procedure: Selective caries removal; Procedure: Selective caries removal with NaOCl
- Pt receiving SCR followed by disinfection with Chlorhexidine (Experimental): The cavity was disinfected with 2% CHX.
  Interventions: Procedure: Selective caries removal; Procedure: Selective caries removal with CHX

INTERVENTIONS:
Procedure: Selective caries removal — Selective caries removal followed by cavity disinfection with NaOCl & CHX in each test group & no cavity disinfection in control group.
Procedure: Selective caries removal with NaOCl — elective caries removal followed by cavity disinfection with NaOCl
  Arms: Pt receiving SCR followed by disinfection with NaOCl
Procedure: Selective caries removal with CHX — elective caries removal followed by cavity disinfection with CHX
  Arms: Pt receiving SCR followed by disinfection with Chlorhexidine

SUMMARY:
To investigate The Effect of Sodium hypochlorite and Chlorhexidine as cavity Disinfectants on the post operative pain and Success of Partial Caries Removal in deep carious lesion with moderate pulpitis in permanent teeth

DETAILED DESCRIPTION:
Study Design: Intervention Research Question : To investigate whether the use of 2% chlorhexidine and 5.25% sodium hypochlorite can improve the clinical and radiographic outcome after partial caries removal in deep carious lesion P (Population) - Mature Permanent Mandibular molars with deep carious lesion involving inner two third of dentine I (Intervention) - - Partial caries removal using 2% chlorhexidine/5.25% sodium hypochlorite as cavity disinfectant..

C (Comparison) - Partial caries removal using saline as cavity disinfectant. O (Outcome) - Assessment of clinical and radiographic success at 12 months follow up.

-To assess incidence and reduction in pain post operatively at every 24 hours till 1 week.

ELIGIBILITY:
Inclusion Criteria:

1. The patient should be ≥18 years of age.
2. Restorable mature permanent 1st and 2nd Mandibular molars with extremely deep caries (≥2/3 dentine involvement)
3. Tooth should give positive response to pulp sensibility testing.
4. Clinical diagnosis of moderate pulpitis.
5. Radiographic finding of periapical index (PAI) score ≤2.
6. Healthy periodontium (probing pocket depth ≤3 mm and mobility within normal limit)

Exclusion Criteria:

Presence of vertical root fracture Presence of root perforations ASA-3 or ASA-4 according to the classification of the American Society of Anesthesiologists) Presence of root resorption Combined endodontic-periodontic lesions. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
Clinical success criteria | 12 months
  No history of spontaneous pain or discomfort except for the initial days after treatment.
  No tenderness to palpation or percussion and the tooth is functional. Normal mobility and probing pocket depth. Soft tissues around tooth are normal with no swelling or sinus tract.
Radiographic success criteria | 12mnths
  No pathosis evident on the radiograph such as root resorption, furcal pathosis or new periapical pathosis.
  Periapical Index score 1 or 2 according to OrstavicKet al.

SECONDARY OUTCOMES:
Pain assesment | 7 days
  Patients will be informed that they may experience pain in the days after treatment and will be instructed to record their pain at 24 h, 2, 3, 4, 5, 6 and 7 days after the treatment, to be submitted after 1 week.
  They will be instructed to use analgesics (Ibuprofen 400 mg every 6-8 h), if needed for pain relief. They will be requested to note down the details of analgesic intake on the pain form regarding the number of doses required, timing of the dose and whether it provided adequate pain relief or not (yes/no) Visual analogue scale (VAS) from 0 to 100 will be used to record preoperative and post -operative pain.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Sanjay Tewari, MDS, Principal Investigator — PGIDS Rohtak
Locations (1):
- Pgids Rohtak, Haryāna, India

IPD SHARING:
Plan to Share IPD: No